CLINICAL TRIAL: NCT01592513
Title: Effect of BIS Monitoring on Propofol Usage During Elective Bronchoscopy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Rabin Medical Center (Other)
Responsible Party: Principal Investigator, Mordechai Kremer, Head of pulmonology institute, Rabin Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: rmc116633CTIL
Record Dates: First submitted 2012-03-14; First posted 2012-05-07 (Estimated); Last update posted 2012-05-07 (Estimated); Status verified 2012-05

CONDITIONS: Pulmonary Diseases
MeSH Terms: conditions — Lung Diseases

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (No Intervention)
- BIS monitor (Experimental): Patients in this group will be monitored by BIS (placement of an electrode over the forehead before sedation).
  Patients in this group will receive propofol (boluses of 10-20 mg) to reach a BIS target value of 80-90.
  Interventions: Device: BIS monitor

INTERVENTIONS:
Device: BIS monitor — BIS is a monitor of anesthetic depth approved by the FDA. It incorporates time-domain, frequency-domain and bi-spectral analysis of the EEG. This analysis is displayed as a dimensionless number between zero (deep anesthesia) and 100 (awake).
  BIS values between 80-90 represent values corresponding to light/moderate sedation.
  BIS is a valuable tool for assessing the depth of sedation and guiding the administration of sedative drugs.
  Other Names: BIS monitor by Covidien - aspectmedical
  Arms: BIS monitor

SUMMARY:
In this research, the investigators will asses the effect of BIS monitoring on propofol usage during elective flexible fiberoptic bronchoscopy.

The investigators will examine whether use of BIS monitor enables reduction of sedative dose during bronchoscopy.

The investigators will also examine whether administration of lower total sedative dose enables prevention of possible complications.

DETAILED DESCRIPTION:
During flexible fiberoptic bronchoscopy (FFP) a narrow optic tube is inserted via the mouth or nose into the airways. This allows direct visualization of the airways as well as taking different samples. In addition, this procedure allows opening of airway obstruction.

Administration of sedation during FFP is important, since this diminishes patient discomfort and body movements. It also lessens the untoward physiologic response to airway manipulation. In addition, patients requiring repeated examinations may refuse if they have suffered an unpleasant experience.

FFP is usually a brief procedure (several minutes up to an hour). Therefore, it is advantageous to use short acting drugs in order to shorten the prolonged post procedural monitoring and allow rapid patient discharge.

Several clinical trials have shown the superiority of propofol over midazolam for sedation during bronchoscopy regarding recovery of alertness, memory & motor function.

Propofol is a sedative-hypnotic with rapid onset and short duration. Using propofol, one can achieve rapid onset of sedation and faster recovery.

Propofol given in boluses of 10-20 mg was found as an effective dose to reach BIS target values.

Awareness is the postoperative recollection of events occurring during general anesthesia.

BIS is a monitor of anesthetic depth approved by the FDA. It incorporates time-domain, frequency-domain and bi-spectral analysis of the EEG. This analysis is displayed as a dimensionless number between zero (deep anesthesia) and 100 (awake).

BIS values between 80-90 represent values corresponding to light/moderate sedation

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years old
* Undergoing flexible fiberoptic bronchoscopy for lung tissue biopsy, airway lavage or opening of airway obstruction.

Exclusion Criteria:

* Patient refusal/ inability to sign informed consent.
* Age under 18 years of age.
* Ventilated patients (via endotracheal tube or tracheostomy).
* Known allergy for one of the anesthetic drugs.
* Patients who suffered a stroke and/or have other neurological diseases.
* Hemodynamically unstable patients (SBP below 90mmHg or above 180mmHg).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2012-04; Primary Completion 2012-08 (Estimated); Study Completion 2012-10 (Estimated)

PRIMARY OUTCOMES:
Total sedative dose in mg. | Duration of flexible fiberoptic bronchoscopy (an average of 30 minutes)

SECONDARY OUTCOMES:
Percentages of patients which developed complications resulting from use of sedatives | Duration of flexible fiberoptic bronchoscopy (an average of 30 minutes) up to 10 minutes after completion of procedure
  The investigators will assess the occurrence of the following complications: hemodynamic instability, hypoxemia, respiratory depression.
Percentages of awareness during flexible fiberoptic bronchoscopy | Duration of flexible fiberoptic bronchoscopy (an average of 30 minutes)

CONTACTS AND LOCATIONS:
Overall Officials: Mordechai Kremer, Prof, Study Director — Head of pulmonolgy institute, Rabin Medical center
Locations (1):
- Rabin Medical center, Petah Tikva, Israel

REFERENCES:
- [Background] Myles PS, Leslie K, McNeil J, Forbes A, Chan MT. Bispectral index monitoring to prevent awareness during anaesthesia: the B-Aware randomised controlled trial. Lancet. 2004 May 29;363(9423):1757-63. doi: 10.1016/S0140-6736(04)16300-9. PMID 15172773
- [Background] Clark G, Licker M, Younossian AB, Soccal PM, Frey JG, Rochat T, Diaper J, Bridevaux PO, Tschopp JM. Titrated sedation with propofol or midazolam for flexible bronchoscopy: a randomised trial. Eur Respir J. 2009 Dec;34(6):1277-83. doi: 10.1183/09031936.00142108. Epub 2009 May 14. PMID 19443532
- [Background] Bould MD, Mahtani DG, Davies R, Roughton M, Hunter DN, Kelleher A. Bispectral index values during elective rigid bronchoscopy: a prospective observational pilot study. Anaesthesia. 2007 May;62(5):438-45. doi: 10.1111/j.1365-2044.2007.04986.x. PMID 17448053
- [Background] Yamamoto S, Igarashi T, Tetsuka K, Endo S. Bispectral index monitoring of midazolam sedation during flexible bronchoscopy. J Bronchology Interv Pulmonol. 2009 Oct;16(4):241-4. doi: 10.1097/LBR.0b013e3181bb781f. PMID 23168586
- [Background] Brice DD, Hetherington RR, Utting JE. A simple study of awareness and dreaming during anaesthesia. Br J Anaesth. 1970 Jun;42(6):535-42. doi: 10.1093/bja/42.6.535. No abstract available. PMID 5423844
- [Result] Carmi U, Kramer MR, Zemtzov D, Rosengarten D, Fruchter O. Propofol safety in bronchoscopy: prospective randomized trial using transcutaneous carbon dioxide tension monitoring. Respiration. 2011;82(6):515-21. doi: 10.1159/000331506. Epub 2011 Sep 16. PMID 21934290
- [Result] Tschopp JM, Purek L, Frey JG, Schnyder JM, Diaper J, Cartier V, Licker M. Titrated sedation with propofol for medical thoracoscopy: a feasibility and safety study. Respiration. 2011;82(5):451-7. doi: 10.1159/000329438. Epub 2011 Oct 13. PMID 21996705
- [Result] Avidan MS, Zhang L, Burnside BA, Finkel KJ, Searleman AC, Selvidge JA, Saager L, Turner MS, Rao S, Bottros M, Hantler C, Jacobsohn E, Evers AS. Anesthesia awareness and the bispectral index. N Engl J Med. 2008 Mar 13;358(11):1097-108. doi: 10.1056/NEJMoa0707361. PMID 18337600
- [Result] I Matot, et al. Sedation in outpatient flexible bronchoscopy: alfentanil-propofol versus Meperidine-Midazolam. Journal of Bronchology & interventional pulmonology 1999; 6:74-77.
- [Result] Mashour GA, Orser BA, Avidan MS. Intraoperative awareness: from neurobiology to clinical practice. Anesthesiology. 2011 May;114(5):1218-33. doi: 10.1097/ALN.0b013e31820fc9b6. PMID 21464699